CLINICAL TRIAL: NCT04900753
Title: Rrisk Factors of Xerostomia (Dry Mouth) After Surgery
Brief Title: Risk Factors Related to Thirst After Surgery
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901244A3
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the risk factors related to xerostomia (dry mouth) after surgery

DETAILED DESCRIPTION:
Dry mouth of postoperative makes the patient feel thirst, and the pain of the lips is cracked. It will also make the sputum thick and sticky, making it difficult for the patient to cough by himself. Especially the elderly may have sputum accumulation and pneumonia. The incidence of dry mouth was 88%, 6-8 hours after abdominal surgery. Initiating the motivation of this study, it is hoped that through research to understand the relevant factors causing dry mouth after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients
2. Elective surgery patients
3. >19 years old patients

Exclusion Criteria:

1. cognitive impairment patients
2. ICU patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: over 19 years old elective surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
To investigate the risk factors related to xerostomia (dry mouth) after surgery | 5 mins
  To investigate the risk factors related to xerostomia (dry mouth) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hsiu-Ling Yang, Taoyuan District, No.5, Fuxing St., Guishan Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No